CLINICAL TRIAL: NCT05431231
Title: Testing the Effectiveness of Two Hospitalization Alternatives Compared to Psychiatric Hospitalization: an Open Comparative Study
Brief Title: Testing the Effectiveness of Two Hospitalization Alternatives Compared to Psychiatric Hospitalization (HOSP-ALT)
Acronym: HOSP-ALT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-19-6555-MW-CTIL
Record Dates: First submitted 2019-11-23; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Questionnaires; Data Collection
Keywords: psychiatric hospitalization; hospitalization alternatives; soteria; online hospitalization

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- psychiatric ward: Adults consenting to treatment, who are admitted in the psychiatric ward at the Sheba Medical Health Center, whose first hospitalization has been up to five years before their current referral.
  Interventions: Diagnostic Test: Outcome Questionnaire-45; Diagnostic Test: Hopkins symptoms checklist - short form; Diagnostic Test: Prodromal Questionnaire - Brief Version; Diagnostic Test: Manchester Short Assessment of Quality; Diagnostic Test: Self-Stigma of Mental Illness Scale; Diagnostic Test: Session Alliance Inventory - for patient; Other: Quality of service/satisfaction questionnaire; Diagnostic Test: Clinical decision-making style; Diagnostic Test: Global Assessment of Functioning Scale; Diagnostic Test: Session Alliance Inventory - for therapist
- Online hospitalization: adults consenting to treatment in their homes, who are found in an acute state that requires hospitalization, whose first hospitalization has been up to five years before their current referral. All the therapeutic treatments, assessment and follow-up meetings that are included in the service are provided online.
  Interventions: Diagnostic Test: Outcome Questionnaire-45; Diagnostic Test: Hopkins symptoms checklist - short form; Diagnostic Test: Prodromal Questionnaire - Brief Version; Diagnostic Test: Manchester Short Assessment of Quality; Diagnostic Test: Self-Stigma of Mental Illness Scale; Diagnostic Test: Session Alliance Inventory - for patient; Other: Quality of service/satisfaction questionnaire; Diagnostic Test: Clinical decision-making style; Diagnostic Test: Global Assessment of Functioning Scale; Diagnostic Test: Session Alliance Inventory - for therapist
- Soteria: adults consenting to treatment in a house in the community, who are found in an acute state that requires hospitalization, whose first hospitalization has been up to five years before their current referral.
  Interventions: Diagnostic Test: Outcome Questionnaire-45; Diagnostic Test: Hopkins symptoms checklist - short form; Diagnostic Test: Prodromal Questionnaire - Brief Version; Diagnostic Test: Manchester Short Assessment of Quality; Diagnostic Test: Self-Stigma of Mental Illness Scale; Diagnostic Test: Session Alliance Inventory - for patient; Other: Quality of service/satisfaction questionnaire; Diagnostic Test: Clinical decision-making style; Diagnostic Test: Global Assessment of Functioning Scale; Diagnostic Test: Session Alliance Inventory - for therapist

INTERVENTIONS:
Diagnostic Test: Outcome Questionnaire-45 — a questionnaire that evaluates the patient's level of distress. The questionnaire was developed by Lambert et al. in 1996 and was translated to Hebrew by Gross, Glasser, Elisha et al. in 2015. The questionnaire is composed of 45 statements that describe emotional states, assessing three main components: subjective discomfort, interpersonal relationships and performance of social roles. The participants are asked to rate how often they have felt the states described by each statement using a five-level Likert scale (0 - never, 4 - almost always). This questionnaire has been used extensively and has showed good internal consistence of 0.93 for its English version and 0.91 for its Hebrew version.
  Other Names: OQ-45
Diagnostic Test: Hopkins symptoms checklist - short form — a questionnaire for assessing symptomatic distress. The questionnaire was developed by Lutz, Tholen, Schürch, and Berking in 2006. It is a short version of the SCL-90-R, that was developed by Derogatis in 1992. The checklist includes 11 items that describe negative feelings and thoughts. Participants are asked to rate the extent to which a given feeling or thought has troubled them in the past week using a four-level Likert scale (1 - not at all, 4 - very much). This tool is highly correlated with the Global Severity Index (r=.91) and has shown high internal consistency.
  Other Names: HSCL-11
Diagnostic Test: Prodromal Questionnaire - Brief Version — a patient questionnaire that assesses the existence of a prodromal state or fully developed psychosis. It was developed by Ising et al. in 2012 and was translated to Hebrew by Koren et al. in 2016. The tool is based on a more extensive questionnaire - PQ-92 - that was developed by Loewy et al. in 2005 - and constitutes an attempt to create an improved shorter version. The PQ-16 includes 16 items that refer to thoughts, feelings and experiences that describe various symptoms, including abnormal perception (9 items), unconventional thinking and paranoia (5 items) and negative symptoms (2 items). For each item, first, the participant is asked to indicate whether he had experienced that phenomenon in the past month, and if he had, he is asked to describe the extent to which the phenomenon had caused him distress, using a four-level Likert scale (0 - no distress, 3 - severe distress). Ising et al. found that Kronbach's α was 0.774 for the whole questionnaire.
  Other Names: PQ-16
Diagnostic Test: Manchester Short Assessment of Quality — a patient questionnaire that assesses quality of life. This questionnaire was developed by Priebe, Huxley, Knight and Evans in 1999. It is based on a longer questionnaire - Lancashire Quality of Life Profile (LQLP) - and was created as an attempt to form an improved shorter version. The questionnaire is composed of two parts: personal details that can change over time and 16 questions that assess objective and subjective quality of life. The objective items are presented as yes or no questions, while regarding the subjective items, participants are asked to describe, using a 7-level Likert scale, the extent to which they are satisfied with their lives. Priebe et al. reported an alpha internal consistency of 0.74.
  Other Names: MANSA
Diagnostic Test: Self-Stigma of Mental Illness Scale — a patient questionnaire that assesses internalized self-stigma. It was developed by Corrigan, Watson, and Barr in 2006. The questionnaire is composed of four dimensions. The questionnaire includes 40 items, 10 items for each dimension. The participant is asked to rate the extent to which he agrees with each item using a 9-level Likert scale. The questionnaire yields four separate scores for each dimension, and each dimension can be administered separately and independently. In the current study, only one 10-item dimension will be administered - the extent to which the participant has internalized stereotypes concerning mental illness. Corrigan et al (2006) reported an internal consistency alpha of 0.81 and a test-retest reliability ratio of 0.82 for this dimension.
  Other Names: SSMIS
Diagnostic Test: Session Alliance Inventory - for patient — this questionnaire has two versions, one for patients and one for the main therapist in the therapeutic team, and its goal is to evaluate the therapist-patient relationship (therapeutic alliance). It is composed of 6 statements that relate to the therapeutic relationship. The participants are asked to rate the extent to which the statements describe their experience accurately using a 7-level Likert scale (1 - does not describe my experience in any way, 7 - describes my experience exactly). In the current study, patients will define who their main therapist is. Falkenstrom et al. reported that in their three tested samples, the alpha coefficients ranged from 0.89 to 0.94.
  Other Names: SAI
Other: Quality of service/satisfaction questionnaire — measured by the quality of service department at Sheba Medical Health Center (or - PROMS, to be decided). Here customer's experience of the online services would be measured as well.
Diagnostic Test: Clinical decision-making style — a questionnaire with two - patient and therapist - versions, meant to evaluate decision making style. It was developed by Puschner, Neumann, Jordan, et al. in 2013. The questionnaire constitutes a modified version of the Autonomy Preference Index (API), which was developed by Ende, Kazis, Ash, & Moskowitz in 1989 for mental health patients. In the current study, only the therapist/psychiatrist version would be administered. The questionnaire is composed of 21 items and yields two components related to clinical decision making: preferences in decision making style and information seeking during decision making. Puschner et al (2013) reported that Kronbach's α coefficient ranged from 0.87 to 0.89.
  Other Names: CDMS
Diagnostic Test: Global Assessment of Functioning Scale — a questionnaire meant to assess the patient's global functioning. It was developed by Jones, Thornicroft, Coffey, & Dunn in 1996. The GAF was used in DSM-IV as the fifth axis of psychiatric evaluation. The therapist is asked to determine for each patient a general score ranging from 10 to 100 to describe his everyday functioning in psychological, social and occupational fields. A score of 10 refers to a state of persistent danger of severely hurting the self or others, and a score of 100 refers to superior functioning in all areas of life. Jones et al. reported that Kronbach's α ranged from 0.74 to 0.76.
  Other Names: GAF
Diagnostic Test: Session Alliance Inventory - for therapist — a questionnaire that has two - patient and therapist - versions, meant to assess the therapist-patient relationship (therapeutic alliance). It was developed by Falkenstrom, Hatcher, Skjulsvik, Larsson, & Holmqvist in 2014. Each questionnaire (patient/therapist) is composed of 6 statements that refer to the therapeutic relationship. The participants are asked to rate the extent to which the statements describe their experience accurately using a 7-level Likert scale (1 - does not describe my experience in any way, 7 - describes my experience exactly). Falkenstrom et al reported that Kronbach's α coefficient ranged from 0.89 to 0.94 for their three tested samples. In the current study, patients will define who their main therapist is.
  Other Names: SAI

SUMMARY:
studies show that many of the people who were hospitalized in psychiatric wards had negative experiences of their stay there. These reports regarding patients' experiences have led in recent years to the development of several hospitalization alternatives that were meant to improve patients' experiences in an acute time in their lives, out of hope that the staying in a familiar and safe place and in one's natural environment will allow better recovery. The current study, is an open comparative study. Testing the effectiveness of two hospitalization alternatives compared to psychiatric hospitalization. First alternative is called Soteria. a house in the community for people who are coping with extreme emotional states. The goal of the house is to allow the coping person to get through the crisis in an open, respectful atmosphere. Second alternative is online home hospitalization. The model uses technological solutions to allow management of effective, integrative treatment for people who are coping with extreme emotional states while they remain in their homes. this model is innovative and has not yet been attempted elsewhere in the world. The goal of the current study is to explore whether there are any differences between hospitalization in psychiatric units, online home hospitalization, and staying in Soteria homes in a series of qualitative, outcome and process measures.

DETAILED DESCRIPTION:
studies show that many of the people who were hospitalized in psychiatric wards had negative experiences. Thus, for example, patients mentioned experiences of uncertainty regarding the treatment that patients received, the rules of the psychiatric ward, length of the hospitalization, nurses' lack of time to interact with patients and even feelings of humiliation. On the other hand, patients noted that the involvement and presence of family and friends during the hospitalization aroused positive feelings. These reports regarding patients' experiences have led in recent years to the development of several hospitalization alternatives that were meant to improve patients' experiences in an acute time in their lives, out of hope that the staying in a familiar and safe place and in one's natural environment will allow better recovery.

One of the first alternatives to inpatient hospitalization that was developed in Israel was Soteria. The Soteria house is a house in the community for people who are coping with extreme emotional states. The therapeutic model is based on a model that was developed in California in the beginning of the seventies by psychiatrist Dr. Loren Mosher and on additional homes in the world that were established upon his inspiration, the oldest one established in Bern, Switzerland in the eighties that is still active today. The goal of the house is to offer an alternative to inpatient psychiatric hospitalization, which would allow the coping person to get through the crisis in an open, respectful atmosphere. In the Soteria house, mental health professionals work in full cooperation with the patient's family and loved ones, with an emphasis on reducing stigma. The house is based on principles of security, open communication, nonjudgmental listening and respectful treatment as necessary conditions for coping and recovery. Every house contains up to 10 residents along with two or three guides, who are usually students who major in therapeutic professions and/or people with a history of receiving psychiatric care ("Peer Specialists"). The daily work in the house is accompanied by a group of professionals that includes a psychiatrist, a psychologist, a social worker and a nurse. In addition, the family-social circle of the resident is offered supportive conversations in the "open dialogue" spirit. The Soteria house has been active in Israel since September 2016 and so far, its effectiveness has not been studied empirically. However, numerous studies of this model were performed in the world and a meta-analysis conducted at 2008 even showed that in the short term, balancing houses decreased the symptomatic level in the same rate as psychiatric wards, while in the long term, they led to higher improvement in patients' quality of life and psycho-social functioning in comparison to inpatient hospitalization units.

Another alternative to inpatient hospitalization that has been applied recently in the Sheba Medical Center at Tel HaShomer is one of online home hospitalization. This setting is an alternative to psychiatric hospitalization that uses technological solutions to allow management of effective, integrative treatment for people who are coping with extreme emotional states while they remain in their homes. The model is based on containment, lack of judgment and cooperation with figures in the community. It was established to try to reduce the damages of acute psychiatric illness, decrease the influences of stigma (that often even leads to avoidance of treatment for a long, crucial period of time) and to significantly improve the experience of the patient and his family. All the therapeutic treatments, assessment and follow-up meetings that are included in the service are provided online. Firstly, the service includes video chats with an interdisciplinary staff that includes a psychiatrist, a psychologist, a social worker, a nurse and an occupational therapist. Secondly, it involves sensors that continuously monitor behavioral data such as medication taking, and physiological data such as sleep, temperature and pulse. Thirdly, it involves reminders to take medication, to participate in follow-up meetings etc. Fourthly, a psychiatric nurse is available to the patient 24/7. Since it is not location dependent, the online service allows the entire staff (psychiatrist, psychologist, social worker) to be there for the patient continuously. Even though this model is innovative and has not yet been attempted elsewhere in the world, it is based on an extensive body of knowledge that demonstrates the effectiveness of online therapy in the treatment of psychological problems.

Despite encouraging data demonstrating the promise of hospitalization alternatives for patients' psychological wellbeing, so far, no studies compared the effectiveness of these models to that of standard psychiatric hospitalization. The goal of the current study is to try to bridge this gap through an open comparative study that examines several measures that are meant to assess the effectiveness of hospitalization alternatives in comparison to psychiatric hospitalization. Specifically, the investigators would like to explore whether there are any differences between hospitalization in psychiatric units, online home hospitalization, and staying in balancing homes in a series of qualitative, outcome and process measures. An emphasis will be made on three main components: symptomatic improvement, improvement in psycho-social functioning and improvement in patient experience. The research hypotheses are as follows:

1. In accordance with previous findings, all three models would lead to similar symptomatic improvement, with no short-term differences.
2. The follow-up measurements would show differences in the quality of life measures; i.e. patients' quality of life and psychological wellbeing are expected to improve significantly in the long-term among patients of both hospitalization alternatives.
3. Differences in patients' satisfaction, compliance and psychosocial functioning are expected, with higher improvement rates in hospitalization alternatives compared to psychiatric hospitalization. However, the investigators do not expect to find any differences between the two hospitalization alternatives.

ELIGIBILITY:
Inclusion Criteria:

* Mental condition requiring psychiatric hospitalization
* History of hospitalizations up to 5 years

Exclusion Criteria:

* A condition requiring forced hospitalization
* poor compliance with treatment
* developmental cognitive disability
* complex organic states including dementia
* patients with severe comorbidity such as substance abuse (drugs, alcohol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults who are found in an acute state that requires hospitalization
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Frequency of repeated hospitalizations after release from each setting. | One year since the release from the hospital or from the alternative settings
  For each subject will be measured, the number of times they have been hospitalized In a psychiatric ward or its alternatives, since the beginning of the study.
Duration of hospitalizations. | One year since the release from the hospital or from the alternative settings
  For each subject will be measured, the number of days that they stayed In a psychiatric ward or its alternatives. In all hospitalizations together (For those who have been hospitalized several times) since the beginning of the study.

SECONDARY OUTCOMES:
Outcome Questionnaire-45 (OQ-45) | The questionnaire will be passed at several time points: Baseline and 6, 12 and 18 months since the release from the hospital or from the alternative settings.
  a questionnaire that evaluates the patient's level of distress. The questionnaire was developed by Lambert et al. in 1996 and was translated to Hebrew by Gross, Glasser, Elisha et al. in 2015. The questionnaire is composed of 45 statements that describe emotional states, assessing three main components: subjective discomfort, interpersonal relationships and performance of social roles. The participants are asked to rate how often they have felt the states described by each statement using a five-level Likert scale (0 - never, 4 - almost always). This questionnaire has been used extensively and has showed good internal consistence of 0.93 for its English version and 0.91 for its Hebrew version.
Hopkins symptoms checklist - short form (HSCL-11) | The questionnaire will be passed at several time points: Baseline and release from the hospital or from the alternative settings and 3 months since the release from the hospital or from the alternative settings.
  a questionnaire for assessing symptomatic distress. The questionnaire was developed by Lutz, Tholen, Schürch, and Berking in 2006. It is a short version of the SCL-90-R, that was developed by Derogatis in 1992. The checklist includes 11 items that describe negative feelings and thoughts. Participants are asked to rate the extent to which a given feeling or thought has troubled them in the past week using a four-level Likert scale (1 - not at all, 4 - very much). This tool is highly correlated with the Global Severity Index (r=.91) and has shown high internal consistency.
Prodromal Questionnaire - Brief Version (PQ-16) | The questionnaire will be passed at several time points: Baseline and release from the hospital or from the alternative settings and 3, 6, 12 and 18 months since the release from the hospital or from the alternative settings.
  a patient questionnaire that assesses the existence of a prodromal state or fully developed psychosis. It was developed by Ising et al. in 2012 and was translated to Hebrew by Koren et al. in 2016. The tool is based on a more extensive questionnaire - PQ-92 - that was developed by Loewy et al. in 2005 - and constitutes an attempt to create an improved shorter version. The PQ-16 includes 16 items that refer to thoughts, feelings and experiences that describe various symptoms, including abnormal perception (9 items), unconventional thinking and paranoia (5 items) and negative symptoms (2 items). For each item, first, the participant is asked to indicate whether he had experienced that phenomenon in the past month, and if he had, he is asked to describe the extent to which the phenomenon had caused him distress, using a four-level Likert scale (0 - no distress, 3 - severe distress). Ising et al. found that Kronbach's α was 0.774 for the whole questionnaire.
Manchester Short Assessment of Quality (MANSA) | The questionnaire will be passed at several time points: Baseline and release from the hospital or from the alternative settings and 3, 6, 12 and 18 months since the release from the hospital or from the alternative settings.
  a patient questionnaire that assesses quality of life. The questionnaire is composed of two parts: personal details that can change over time (education, occupational state, family state and income) and 16 questions that assess objective (4 items) and subjective (12 items) quality of life. The objective items are presented as yes or no questions, while regarding the subjective items, participants are asked to describe, using a 7-level Likert scale, the extent to which they are satisfied with their lives.
Self-Stigma of Mental Illness Scale (SSMIS) | The questionnaire will be passed at several time points: Baseline and release from the hospital or from the alternative settings and 3, 6, 12 and 18 months since the release from the hospital or from the alternative settings.
  a patient questionnaire that assesses internalized self-stigma. The questionnaire is composed of four parts/dimensions: level of awareness of common stereotypes concerning others who suffer from mental illness, level of agreement with stereotypes concerning others who suffer from mental illness, the extent to which the participant has internalized these stereotypes, and the influence of the stereotypes' internalization on the participant's self-esteem. The questionnaire includes 40 items, 10 items for each dimension. each dimension can be administered separately and independently. In the current study, only one 10-item dimension will be administered - the extent to which the participant has internalized stereotypes concerning mental illness.
Session Alliance Inventory (SAI) - To the patient | The questionnaire will be passed at several time points: Baseline and release from the hospital or from the alternative settings and 3, 6, 12 and 18 months since the release from the hospital or from the alternative settings.
  this questionnaire has two versions, one for patients and one for the main therapist in the therapeutic team, and its goal is to evaluate the therapist-patient relationship (therapeutic alliance). It is composed of 6 statements that relate to the therapeutic relationship. The participants are asked to rate the extent to which the statements describe their experience accurately using a 7-level Likert scale (1 - does not describe my experience in any way, 7 - describes my experience exactly). In the current study, patients will define who their main therapist is. Falkenstrom et al. reported that in their three tested samples, the alpha coefficients ranged from 0.89 to 0.94.
Quality of service/satisfaction questionnaire | The questionnaire will be passed at several time points: Baseline and release from the hospital or from the alternative settings.
  measured by the quality of service department at Sheba Medical Health Center (or - PROMS, to be decided). Here customer's experience of the online services would be measured as well.
Clinical decision-making style (CDMS) | Baseline
  a questionnaire with two - patient and therapist - versions, meant to evaluate decision making style. In the current study, only the therapist/psychiatrist version would be administered once, in the beginning of the study, regarding all patients in general. The questionnaire is composed of 21 items and yields two components related to clinical decision making: preferences in decision making style and information seeking during decision making.
Global Assessment of Functioning Scale (GAF) | The questionnaire will be passed at several time points: Baseline and release from the hospital or from the alternative settings and 3, 6, 12 and 18 months since the release from the hospital or from the alternative settings.
  a questionnaire meant to assess the patient's global functioning. It was developed by Jones, Thornicroft, Coffey, & Dunn in 1996. The GAF was used in DSM-IV as the fifth axis of psychiatric evaluation. The therapist is asked to determine for each patient a general score ranging from 10 to 100 to describe his everyday functioning in psychological, social and occupational fields. A score of 10 refers to a state of persistent danger of severely hurting the self or others, and a score of 100 refers to superior functioning in all areas of life. Jones et al. reported that Kronbach's α ranged from 0.74 to 0.76.
Session Alliance Inventory (SAI) - To the therapist | The questionnaire will be passed at several time points: Baseline and release from the hospital or from the alternative settings and 3, 6, 12 and 18 months since the release from the hospital or from the alternative settings.
  a questionnaire that has two - patient and therapist - versions, meant to assess the therapist-patient relationship (therapeutic alliance). It was developed by Falkenstrom, Hatcher, Skjulsvik, Larsson, & Holmqvist in 2014. Each questionnaire (patient/therapist) is composed of 6 statements that refer to the therapeutic relationship. The participants are asked to rate the extent to which the statements describe their experience accurately using a 7-level Likert scale (1 - does not describe my experience in any way, 7 - describes my experience exactly). Falkenstrom et al. reported that Kronbach's α coefficient ranged from 0.89 to 0.94 for their three tested samples. In the current study, patients will define who their main therapist is.

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Soteria Home for Women, Jerusalem
  - Soteria Home for Men, Jerusalem
  - Soteria Home in the Sharon, Kfar Yona
  - Sheba Medical Center, Psychiatry Department, Ramat Gan